CLINICAL TRIAL: NCT05039619
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Obinutuzumab in Adolescent Patients With Active Class III or IV Lupus Nephritis, Including an Evaluation of Open Label Safety and PK in a Cohort of Pediatric Patients (Aged 5 to < 12)
Brief Title: A Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Obinutuzumab in Adolescents With Active Class III or IV Lupus Nephritis and the Safety and PK of Obinutuzumab in Pediatric Participants
Acronym: POSTERITY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA42985; 2021-000097-29 (EudraCT Number); 2023-505825-15-00 (Other: EU CT Number)
Record Dates: First submitted 2021-09-01; First posted 2021-09-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — obinutuzumab; Mycophenolic Acid; Acetaminophen; Diphenhydramine; Methylprednisolone; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Blinded Obinutuzumab (Experimental): Participants will receive obinutuzumab 1000 milligrams (mg) intravenous (IV) infusions on Day 1, Day 14, Week 24, Week 26 and Week 52. Participants with a body weight of 45 kg or more will receive the 1000 mg dose. Participants with a body weight below 45 kg will receive a weight adjusted dose of 20 mg/kilogram (kg).
  Interventions: Drug: Obinutuzumab; Drug: Mycophenolate Mofetil; Drug: Acetaminophen/paracetamol; Drug: Diphenhydramine hydrochloride (HCl); Drug: Methylprednisolone; Drug: Prednisone
- Placebo (Placebo Comparator): Placebo participants will receive obinutuzumab matched placebo on Day 1, Day 14, Week 24, Week 26 and Week 52.
  Interventions: Drug: Placebo; Drug: Mycophenolate Mofetil; Drug: Acetaminophen/paracetamol; Drug: Diphenhydramine hydrochloride (HCl); Drug: Methylprednisolone; Drug: Prednisone
- Open-Label Obinutuzumab (Experimental): Younger participants aged 5 to <12 will receive obinutuzumab 1000 mg IV infusions on Days 1, 14, Week 24, Week 26 and Week 52.
  Interventions: Drug: Obinutuzumab; Drug: Mycophenolate Mofetil; Drug: Acetaminophen/paracetamol; Drug: Diphenhydramine hydrochloride (HCl); Drug: Methylprednisolone; Drug: Prednisone

INTERVENTIONS:
Drug: Obinutuzumab — Obinutuzumab will be administered by IV infusion at a dose of 1000 mg on Day 1, Day 14, Week 24, Week 26 and Week 52.
  Other Names: Gazyva
  Arms: Blinded Obinutuzumab; Open-Label Obinutuzumab
Drug: Placebo — Placebo matching obinutuzumab will be administered by IV on Day 1, Day 14, Week 24, Week 26 and Week 52.
  Arms: Placebo
Drug: Mycophenolate Mofetil — Mycophenolate Mofetil (MMF) will be taken by home administration orally at a target dose of 1200 mg/m^2/day to a maximum of 2.5g/day from baseline (Day 1) onwards.
Drug: Acetaminophen/paracetamol — Acetaminophen 1000 mg will be administered as pre-medication prior to infusions.
Drug: Diphenhydramine hydrochloride (HCl) — Diphenhydramine HCl 50 mg will be administered as pre-medication prior to infusions.
Drug: Methylprednisolone — Methylprednisolone 80 mg IV will be administered as pre-medication prior to infusions.
Drug: Prednisone — Oral prednisone or equivalent corticosteroid will be taken by home administration daily to a maximum dose of 60mg/day followed by a guided taper to 5mg/day or less by Week 24.

SUMMARY:
This phase II, randomized, double-blind, placebo-controlled study is designed to evaluate the safety, efficacy and pharmacokinetics (PK) of obinutuzumab in adolescent participants (AP) aged 12 to less than 18 with biopsy-confirmed proliferative lupus nephritis (LN). It will also evaluate open label safety and PK of obinutuzumab in pediatric participants (PP), aged 5 to <12 with LN.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are age 12 to <18 years at the time of randomization
* Participants who are age 5 to <12 years (younger participant cohort) at the time of randomization once recruitment is open. (Investigators will be notified by the Sponsor when recruitment is open to this younger population)
* International Society of Nephrology and the Renal Pathology Society (ISN/RPS) 2003 Class III or IV active LN demonstrated on renal biopsy performed in the 12 months prior to or during screening
* Class V disease may be present in addition to Class III or IV LN, but participants with isolated Class V disease are not eligible
* Diagnosis of SLE according to the Systemic Lupus International Collaborating Clinics (SLICC) 2012 criteria
* Significant proteinuria defined by a UPCR above > 0.5 based on a first-morning void (FMV) collection at screening
* During the 12 months prior to or during screening, all participants must have received at least one dose of pulse-range IV methylprednisolone (typically 30 mg/kg, maximum of 1000 mg per dose) or equivalent for the treatment of the current episode of active LN.

Exclusion Criteria:

* Severe, active central nervous system (CNS) SLE, including retinitis, poorly controlled seizure disorder, acute confusional state, myelitis, stroke, cerebellar ataxia, or dementia
* Sclerosis in >50% of glomeruli on renal biopsy
* Purely chronic Class III(c) or Class IV(c) disease on renal biopsy, defined as the absence of any active lesions
* Presence of rapidly progressive glomerulonephritis
* Pure Class V LN
* Intolerance or contraindication to study therapies
* Active infection of any kind (excluding fungal infection of nail beds) or any major episode of infection requiring hospitalization or treatment with IV anti-infective medications within 4 weeks prior to screening, or completion of oral anti-infectives within 2 weeks prior to randomization
* History of or currently active primary or secondary immunodeficiency, including known history of HIV infection and other severe Immunodeficiency blood disorders
* History of serious recurrent or chronic infection
* History of or current cancer, including solid tumors, hematological malignancies, and carcinoma in situ (except basal cell carcinoma and squamous cell carcinoma of the skin that have been excised and cured) within the past 5 years
* Significant or uncontrolled concomitant medical disease which, in the investigator's opinion, would preclude participant participation
* Currently active alcohol or drug abuse or history of alcohol or drug abuse

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2029-09-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve a Complete Renal Response (CRR) (AP) | Week 76
  CRR is defined as achievement of all of the following:
  * Urinary protein-to-creatinine ratio (UPCR) <0.5 g/g
  * Estimated Glomerular Filtration Rate (eGFR) >=85% of baseline
  * No occurrence of intercurrent events
Percentage of Participants with Adverse Events (PP) | Baseline to Week 76

SECONDARY OUTCOMES:
Percentage of Participants Achieving a CRR (AP) | Weeks 24 and 52
Percentage of Participants who Achieve CRR with Successful Prednisone Taper (AP) | Week 76
Percentage of Participants who Achieve a PRR (AP) | Week 76
Percentage of Participants Achieving an Overall Response (CRR or PRR) (AP) | Weeks 24, 52, and 76
  PRR is defined as:
  achievement of all of the following:
  * >=50% reduction in urinary protein-to-creatinine ratio (UPCR) from baseline
  * UPCR < 1 g/g (or < 3 g/g if the baseline UPCR was >=3 g/g)
  * eGFR >=85% of baseline
  * No occurrence of intercurrent events
Change in UPCR (AP) | Baseline to Week 76
Change in eGFR (AP) | Baseline to Week 76
Time to Onset of CRR over the Course of 76 weeks (AP) | Up to Week 76
Percentage of Participants who Experience Treatment Failure (AP) | Week 12 to Week 76
Change in anti-dsDNA titers (AP) | Baseline to Week 76
Change in C3 Complement Levels (AP) | Baseline to Week 76
Change in C4 Complement Levels (AP) | Baseline to Week 76
Percentage of Participants with Adverse Events According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 (AP) | Baseline to Week 76
Serum Concentrations of Obinutuzumab (AP) | Baseline to Week 76
Percentage of Participants Achieving B-cell Depletion (AP) | Baseline, Weeks 4, 24, 52 and 76
Change in Pediatric Quality of Life Inventory-Multidimensional Fatigue Scale (PedsQL)-Fatigue Total Score (AP) | Baseline to Week 76
Change in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) (AP) | Baseline to Week 76
Change from Baseline in Child Health Questionnaire-Parent Form 28 (CHQ-PF28) Domain Scores (AP) | Baseline to Week 76
Percentage of Participants with Anti-drug Antibodies (ADA) (AP) | Weeks 0, 24, 52 and 76
Relationship Between ADA Status and Percentage of Participants Achieving a CRR (AP) | Weeks 24, 52 and 76
Percentage of Participants Achieving a CRR (PP) | Week 76
Percentage of Participants Achieving an Overall Response (PP) | Week 76
  PRR is defined as achievement of all of the following:
  * >=50% reduction in UPCR from baseline
  * UPCR < 1 g/g (or < 3 g/g if the baseline UPCR was >=3 g/g)
  * eGFR >=85% of baseline
  * No occurrence of intercurrent events
Percentage of Participants who Achieve CRR with Successful Prednisone Taper (PP) | Week 76
Change in eGFR (PP) | Baseline to Week 76
Percentage of Participants Achieving B-cell Depletion (PP) | Baseline, Weeks 4, 24, 52 and 76
Percentage of Participants with ADAs (PP) | Weeks 0, 24, 52 and 76
Change in anti-dsDNA titers (PP) | Baseline to Week 76

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (42):
- United States (11):
  - Loma Linda University health, Loma Linda, California
  - UCSF Benioff Childrens Hospital, San Francisco, California
  - Children's Hospital Colorado, Anchutz Medical Campus, Aurora, Colorado
  - Emory Children's Center, Atlanta, Georgia
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Louisiana State University, Shreveport, Louisiana
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cohen Children's Medical Center of New York, Queens, New York
  - Cincinnati Childrens Hospital, Cincinnati, Ohio
  - Chldren?s Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Arthritis Center, El Paso, Texas
- Brazil (4):
  - Ser Servicos Especializados Em Reumatologia, Salvador, Estado de Bahia
  - Centro de Pesquisa São Lucas, Campinas, São Paulo
  - Hospital das Clinicas - FMUSP, São Paulo, São Paulo
  - Universidade Federal de Sao Paulo - UNIFES, São Paulo
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - Hospital Sainte-Justine, Montreal, Quebec
- France (4):
  - CH de Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Robert Debré, Paris
  - Hop Necker Enfants Malades, Paris
  - CHU de Toulouse - Hôpital des Enfants, Toulouse
- Italy (3):
  - Ospedale Pediatrico Bambino Gesu, Rome, Lazio
  - IRCCS G. Gaslini, Genoa, Liguria
  - Clinica Pediatrica II De Marchi, Milan, Lombardy
- Mexico (3):
  - CREA Hospital Mexico Americano, Guadalajara, Jalisco
  - Clinstile S.A de C.V., Mexico City, Mexico CITY (federal District)
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
- Peru (2):
  - Instituto de Ginecología y Reproducción, Lima
  - Clinica El Golf, San Isidro
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szpital Specjalistyczny dla Dzieci i Doroslych, Torun
- Saint-Petersburg State, St-peterburg, Sankt-Peterburg, Russia
- South Africa (3):
  - Red Cross War Memorial Children?s Hospital, Cape Town
  - Groote Schuur Hospital, Cape Town
  - Panaroma Medical Center, Panorama
- Spain (4):
  - Hospital Sant Joan De Deu, Esplugas de Llobregat, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Hospital de La Paz, Madrid
  - Hospital Universitario la Fe: Servicio de Reumatologia Pediatrica, Valencia
- United Kingdom (3):
  - Royal Hospital For Children, Glasgow
  - Alder Hey Childrens Hospital, Liverpool
  - Great Ormond Street Hospital for Children, London

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Dossier C, Bonneric S, Baudouin V, Kwon T, Prim B, Cambier A, Couderc A, Moreau C, Deschenes G, Hogan J. Obinutuzumab in Frequently Relapsing and Steroid-Dependent Nephrotic Syndrome in Children. Clin J Am Soc Nephrol. 2023 Dec 1;18(12):1555-1562. doi: 10.2215/CJN.0000000000000288. Epub 2023 Sep 6. PMID 37678236